CLINICAL TRIAL: NCT03940261
Title: Physiological Benefits of High-intensity Interval Training for Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Parkinson Society Canada (Other); YMCA (Other)
Responsible Party: Principal Investigator, Philip Millar, Assistant Professor, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-08-001
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Exercise Training
Keywords: High intensity interval training
MeSH Terms: conditions — Parkinson Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to 10 weeks of either high intensity interval training or continuous moderate intensity training. Training will be conducted in parallel.
Who Masked: Outcomes Assessor
Masking Description: The collection of study outcomes will be completed by individuals blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (Experimental)
  Interventions: Other: High Intensity Interval Training
- Continuous Moderate Intensity Training (Active Comparator)
  Interventions: Other: Continuous Moderate Intensity Training

INTERVENTIONS:
Other: High Intensity Interval Training — Participants will complete exercise training 3x/week for 10 weeks. Exercise will consist of 10, 1-minute cycling intervals at 90% of peak power output, each separated by 1-min at 10% peak power output.
  Arms: High Intensity Interval Training
Other: Continuous Moderate Intensity Training — Participants will complete exercise training 3x/week for 10 weeks. Exercise will consist of 30-50 minutes of cycling at 60% peak power output.
  Arms: Continuous Moderate Intensity Training

SUMMARY:
Aerobic exercise is recommended for individuals with Parkinson's disease (PD) and can improve quality of life, both physically and mentally. The most efficacious program to achieve these exercise benefits is unknown. Recently, high-intensity interval training (HIIT) has been shown to be safe and more effective in many high-risk populations with limited exercise tolerance. Shorter bouts of exercise are likely better tolerated in PD due to difficulty sustaining muscle contractions. The goal of this project is to determine whether HIIT produces superior cardiorespiratory, neuromuscular, biomechanical, and clinical adaptations than conventional continuous moderate intensity training (CMIT) in PD.

DETAILED DESCRIPTION:
The specific research aims are to compare, in PD, the effects of HIIT or CMIT on: 1) maximal exercise capacity; 2) neural and non-neural factors contributing to muscle strength, power and fatigability; 3) biomechanical measures of postural stability and gait; and 4) Clinical markers (Mini-BESTest and Unified Parkinson's Disease Rating Scale (UPDRS)). The investigators hypothesize that, HIIT will produce greater improvements in: 1) exercise capacity; 2) muscle strength, power and reduced fatigability; 3) stability and gait velocity; and 4) clinical markers.

Methods: This pilot project will involve a randomized trial of 30 individuals with PD comparing the effects of HIIT and CMIT. Training will be completed thrice weekly for 10 weeks. Participants will include men and women between 50-85 years of age, who are able to stand unsupported for 1 min, walk 18m without use of an aid, and mount a stationary bike. Participants will be randomized to either HIIT (10, 1-minute cycling intervals at 90% of peak power output, each separated by 1-min at 10% peak power output) or CMIT (30-50min cycling at 60% of peak power output). Participants will undergo the following pre- and post-training assessments: Cardiovascular testing will examine hemodynamic and efferent muscle sympathetic responses to static handgrip exercise and post-exercise circulatory occlusion; Neuromuscular testing will examine muscle activity (electromyography) during voluntary and electrically stimulated contractions of the knee extensors; Biomechanical testing will examine whole-body stability, gait, and balance patterns; and Clinical risk assessments (Mini-BESTest and UPDRS).

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 45-85 years of age
* Clinical diagnosis of Parkinson disease
* Able to stand unsupported for 1 minute
* Able to walk 18 metres without aid
* Able to mount a stationary bike

Exclusion Criteria:

* History of dementia
* History of stroke
* Type 1 diabetes
* Autonomic neuropathy
* Currently involved in formal exercise training (>3 day per week).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | Change from baseline following 10 weeks of aerobic exercise training
  VO2 max

SECONDARY OUTCOMES:
Handgrip strength | Change from baseline following 10 weeks of aerobic exercise training
  Maximal handgrip strength
Blood Pressure | Change from baseline following 10 weeks of aerobic exercise training
  Systolic and Diastolic Blood Pressure
Heart Rate | Change from baseline following 10 weeks of aerobic exercise training
  Cardiovascular measure
Mini-Balance Evaluation Systems Test (Mini-BESTest) | Change from baseline following 10 weeks of aerobic exercise training
  Rating scale consisting of 14 items that are each scored from 0-2, where "0" indicates the lowest level of function and "2" the highest level of function. The test has a maximum score of 28 points.
Unified Parkinson's Disease Rating Scale (UPDRS) | Change from baseline following 10 weeks of aerobic exercise training
  We will use the rating scale to examine 3 segments. 1) MENTATION, BEHAVIOR AND MOOD - 4 questions scored between "0" and "4"; 2) ACTIVITIES OF DAILY LIVING - 13 questions scored between "0" and "4"; and 3) MOTOR EXAMINATION - 14 questions scored between "0" and "4". In each case, a score of "0" indicates normal responses.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Millar, PhD, Principal Investigator — University of Guelph
Locations (1):
- University of Guelph, Guelph, Ontario, Canada